CLINICAL TRIAL: NCT03017625
Title: Platelet Activation and Responsiveness in Patients With Acute Exacerbations of Chronic Obstructive Pulmonary Disease (AE-COPD)
Brief Title: Platelet Activation and Reactivity in Acute Exacerbations of COPD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-2847
Record Dates: First submitted 2016-12-12; First posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: COPD Exacerbation
Keywords: COPD; Cardiovascular Disease; Platelets; Inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cardiovascular Diseases; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood, plasma
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Blood is drawn — Blood analyses

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is known for development of severe cardiovascular co-morbidities. Systemic inflammation during acute exacerbations of COPD (AE-COPD) is thought to play a role in development of cardiovascular disease. Platelets contribute to acute cardiovascular events and atherosclerosis. When platelets are activated, they form complexes with monocytes. These platelet-monocyte complexes (PMCs) are an early process in atherothrombosis and promote inflammation. In COPD, platelet function in AE-COPD is scarcely studied. This study aims to address this gap by investigating platelet function and coagulation in patients with AE-COPD and after convalescence.

ELIGIBILITY:
Inclusion Criteria:

* >40 years
* Spirometry confirmed diagnosis of COPD (i.e. post-bronchodilator FEV1/FVC < 70% and less than 12% on reversibility testing< Lower limit of normal (LLN))
* ≥10 pack years of smoking

Exclusion Criteria:

* Use of anti-coagulation or other platelet function inhibitors
* Asthma
* Chronic inflammatory diseases, for example rheumatoid arthritis, psoriasis, inflammatory bowel diseases , systemic lupus erythematous (SLE)
* Malignancies

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an acute exacerbation of COPD as defined by the Anthonisen criteria
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-01; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Platelet activation: platelet expression of CD62P (P-selectin) and fibrinogen binding at baseline and upon ex vivo stimulation. | Measured at presentation with an AE-COPD and after 8 weeks

SECONDARY OUTCOMES:
Platelet-monocyte interaction (CD14 cells positive for CD61) | Measured at presentation with an AE-COPD and after 8 weeks
Monocyte activation (CD11b expression on CD14 positive cells) | Measured at presentation with an AE-COPD and after 8 weeks
Tissue factor triggered thrombin generation capacity | Measured at presentation with an AE-COPD and after 8 weeks
Plasma markers: Interleukin-6, Interleukin-8, high sensitive-CRP, soluble P-selectin, soluble Fibrinogen, D-dimer | Measured at presentation with an AE-COPD and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne F Heijdra, Md, PhD, Principal Investigator — Radboud University Medical Center